CLINICAL TRIAL: NCT04047940
Title: A Relative Bioavailability Study of Three LY900020 Tablet Formulations in Healthy Chinese Subjects
Brief Title: A Study of LY900020 in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16968; I9J-MC-DIPA (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03-01

CONDITIONS: Healthy
MeSH Terms: interventions — Atorvastatin; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- LY900020 Formulation 1 (Experimental): LY900020 Formulation 1 administered orally
  Interventions: Drug: LY900020
- LY900020 Formulation 2 (Experimental): LY900020 Formulation 2 administered orally
  Interventions: Drug: LY900020
- LY900020 Formulation 3 (Experimental): LY900020 Formulation 3 administered orally
  Interventions: Drug: LY900020
- Reference Drugs (Active Comparator): Metformin XR, atorvastatin, and valsartan administered orally
  Interventions: Drug: Metformin XR; Drug: Atorvastatin; Drug: Valsartan

INTERVENTIONS:
Drug: LY900020 — Administered orally
  Arms: LY900020 Formulation 1; LY900020 Formulation 2; LY900020 Formulation 3
Drug: Metformin XR — Administered orally
  Arms: Reference Drugs
Drug: Atorvastatin — Administered orally
  Arms: Reference Drugs
Drug: Valsartan — Administered orally
  Arms: Reference Drugs

SUMMARY:
This study will evaluate three new formulations of LY900020; a fixed dose, combination drug developed for people with type 2 diabetes mellitus. The study will be conducted in healthy participants to investigate the effect of different tablet formulations on the amount of LY900020 in the bloodstream. Side effects and tolerability will be documented. The study will last about 10 weeks for each participant, including screening and follow up. Screening is required within 28 days prior to entering the study.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy male or a female (not pregnant and agreeable to take birth control measures until study completion)
* Have a body mass index (BMI) of 18.5 to 35 kilogram per square meter (kg/m²), inclusive, at screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), blood and urine laboratory test results that are acceptable for the study

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Had blood loss of more than 400 milliliters (mL) within the last 3 months

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY900020 | Predose through 72 hours postdose on Day 4 in each study arm
  PK: AUC of LY900020
PK: Maximum Observed Drug Concentration (Cmax) of LY900020 | Predose through 72 hours postdose on Day 4 in each study arm
  PK: Cmax of LY900020

SECONDARY OUTCOMES:
PK: Time to Maximum Observed Drug Concentration (tmax) of LY900020 | Predose through 72 hours postdose on Day 4 in each study arm
  PK: Tmax of LY900020

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No